CLINICAL TRIAL: NCT00005240
Title: Correlates of Nonadherence to Hypertension Treatment in an Inner-City Minority Population
Brief Title: Epidemiology of Hypertensive Emergency
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CUMC ID unknown (1121); R01HL038260 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To test the hypotheses that hypertensive emergency was associated with non-compliance with antihypertensive medication, low level of contact with the medical care system, and alcohol abuse and cigarette smoking. Also, to describe the clinical characteristics of patients hospitalized with hypertensive emergency including morbidity, mortality, and cost, and the extent to which hypertensive emergency occured among previously diagnosed and treated hypertensives.

DETAILED DESCRIPTION:
BACKGROUND:

While less frequent than in the era before effective treatment for hypertension, hypertensive emergency remains a relatively common cause of hospital admission in some sub-populations. In 1989, hypertensive emergency accounted for approximately 60 admissions per year to the Medical Service at Presbyterian Hospital, and a somewhat higher proportion of intensive care unit admissions and utilization. The importance of hypertensive emergency may have been underestimated because the International Classification of Diseases discharge codes included only malignant hypertension, a severe form comprising only about half of the admissions for hypertensive emergency. There had been almost no epidemiologic studies of hypertensive emergency since 1969, and very little was known about risk factors.

DESIGN NARRATIVE:

A matched case-control study design was used. Cases were obtained from admissions to the Medical Service at Presbyterian Hospital. Morbidity and mortality data were obtained by follow-up of the case series.

ELIGIBILITY:
Inclusion criteria

1. Patients admitted in the emergency room and for the medical and surgical services at the Presbyterian Hospital and Harlem Hospital Center in New York City

* patients with incidents of hypertensive emergency or hypertensive urgency
* hypertensive patients with other acute conditions who were admitted to the hospital or were treated in the emergency room and released

Exclusion criteria

1. Under 21 years of age
2. Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were enrolled in a case-control study of hypertensive emergency and urgency. Cases were patients with incidents of hypertensive emergency or hypertensive urgency, and controls were hypertensive patients with other acute conditions who were admitted to the hospital or were treated in the emergency room and released.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 1989-10; Primary Completion 1991-06 (Actual); Study Completion 1992-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shea, MD, Principal Investigator — Hamilton Southworth Professor of Medicine and Professor of Epide, Dept of Medicine General Medicine
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Shea S, Misra D, Ehrlich MH, Field L, Francis CK. Correlates of nonadherence to hypertension treatment in an inner-city minority population. Am J Public Health. 1992 Dec;82(12):1607-12. doi: 10.2105/ajph.82.12.1607. PMID 1456334
- [Background] Shea S, Misra D, Ehrlich MH, Field L, Francis CK. Predisposing factors for severe, uncontrolled hypertension in an inner-city minority population. N Engl J Med. 1992 Sep 10;327(11):776-81. doi: 10.1056/NEJM199209103271107. PMID 1501654